CLINICAL TRIAL: NCT05937854
Title: Effect of PDE5 Inhibitor on Respiratory Symptoms in COPD Complicated by Pulmonary Hypertension
Brief Title: Breathe Easier With Tadalafil Therapy for Dyspnea in COPD-PH
Acronym: BETTER COPD-PH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Atlanta VA Medical Center (U.S. Federal Agency); VA Eastern Colorado Health Care System (U.S. Federal Agency); VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PULM-002-22F; I01CX002543 (NIH)
Record Dates: First submitted 2023-06-27; First posted 2023-07-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Hypertension; Dyspnea
Keywords: COPD; cigarette smoke; lung; echocardiography; chest CT; physical activity; spirometry; dyspnea; clinically important deterioration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary; Dyspnea; Cigarette Smoking; Motor Activity | interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: double blind placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be assigned a study code
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Encapsulated placebo one or 2 encapsulated tablets po QD
  Interventions: Drug: Placebo
- tadalafil (Active Comparator): one or 2 encapsulated tablets of encapsulated tadalafil (20MG) po QD
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — one or 2 encapsulated tablets of encapsulated tadalafil (20MG) po QD
  Other Names: Adcirca, Cialis
  Arms: tadalafil
Drug: Placebo — one or two encapsulated tablets of placebo po QD
  Arms: Placebo

SUMMARY:
The investigators will study whether the drug tadalafil improves shortness of breath in 126 Veterans with Chronic Obstructive Pulmonary Disease (COPD) and high blood pressure in the lungs. The investigators will also assess whether tadalafil improves quality of life, home daily physical activity, exercise endurance, the frequency of acute flares of COPD, blood pressure in the lungs, and lung function. Veterans who enroll in the trial will be allocated by chance to either active tadalafil or an inactive identical capsule (placebo). Neither the Veteran nor the investigator will know whether the Veteran is taking tadalafil or placebo. Veterans will be followed closely in clinic or by telephone at 1, 2, 3, 4, 5, and 6 months, with attention to side effects and safety. At 1,3, and 6 months the investigators will repeat the questionnaires and testing of blood pressures in the lung and lung function. The investigators anticipate that the results of this study will determine whether tadalafil improves shortness of breath when added to usual medications for COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is the fourth leading cause of death in the US and is common among Veterans. Dyspnea, a debilitating symptom of COPD, dramatically worsens health related quality of life, is associated with a reduction in daily physical activity and greater health care utilization and is more closely associated with survival than severity of airflow limitation. Thus, it is important to have effective treatments that reduce dyspnea for Veterans with COPD. Pulmonary hypertension (PH) is a common complication of COPD that is associated with severe dyspnea, more frequent acute exacerbations of COPD, and increased mortality. There are multiple causes of PH associated with COPD (COPD-PH), including decreased bioavailable levels of the vasodilator nitric oxide (NO). Phosphodiesterase type-5 inhibitor (PDE-5i) therapy restores NO signaling and improves cardiopulmonary hemodynamics and dyspnea among patients with Pulmonary Arterial Hypertension. However, studies of PDE-5i medications in COPD-PH have shown conflicting results due to differing doses or durations of therapy and differing definitions of PH. In a prior study (ClinicalTrials.gov.identifier: NCT01862536), the investigators investigated the effects of up to 12 months of oral PDE-5i therapy with tadalafil on 6 minute walk distance (6MWD), a measure of exercise capacity in Veterans with COPD-PH, in a multi-center randomized placebo-controlled trial funded by the Department of Veterans Affairs. While tadalafil did not change 6MWD at 6 and 12 months (the primary outcome), the treatment group experienced changes in important secondary outcomes, with clinically meaningful improvement in patient-reported dyspnea and COPD-related health related quality of life after 6 months of therapy. Additionally, over 6 months, dyspnea worsened in the placebo group, and patients receiving PDE-5i therapy suffered fewer exacerbations. A limitation of this study was its small sample size. Given the importance of mitigating dyspnea among patients with COPD, the investigators will assess the effect of maximally tolerated therapy with tadalafil specifically on dyspnea powered as a primary outcome. In 126 participants with COPD-PH (63 treatment and 63 placebo) receiving usual clinical care for COPD, the investigators propose to evaluate effects of tadalafil on dyspnea among patients with COPD-PH in a prospective, double-blind, placebo-controlled clinical trial.

Aim 1: As primary outcome, the investigators will determine whether 6 months of daily oral tadalafil is more effective than placebo in reducing severity of patient-reported dyspnea, assessed by the University of California-San Diego Shortness of Breath Questionnaire (UCSD-SOBQ), in Veterans with COPD-PH. The investigators hypothesize that patients receiving tadalafil will report less dyspnea than those receiving placebo.

Aim 2: As a secondary outcome, the investigators will determine the effectiveness of tadalafil therapy on physical activity, assessed by objective daily step count, and functional capacity, assessed by 6MWD. The investigators hypothesize that patients on tadalafil therapy will have improved physical activity and functional capacity.

Aim 3: As a secondary outcome, the investigators will also assess the effects of tadalafil therapy on time to clinically important deterioration, a validated composite outcome defined as increase > 4U in the total health-related quality of life (St. George's Respiratory Questionnaire, SGRQ), decreased FEV1 of > 100ml, or moderate-severe acute exacerbations of COPD. The investigators hypothesize that Veterans with COPD-PH receiving tadalafil will be less likely to have clinically important deterioration.

Aim 4: In exploratory analyses, the investigators will assess whether changes in noninvasive measures of PH (CT scan, cardiac echo) are associated with changes in dyspnea. The investigators hypothesize that patients receiving tadalafil will have decreased PA/A ratio on CT scan, and decreased ePASP on echocardiography.

This study may provide evidence for a new therapy for dyspnea in COPD complicated by PH.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with COPD, defined as airflow limitation with post-bronchodilator obstruction on baseline visit spirometry, identified by FEV1/FVC < 70% or < the lower limit of normal (5th percentile of a normal population based on Global Lung Function Initiative reference equations), OR any emphysema on chest CT noted in a clinical radiology report confirmed by study investigator review.
2. Eligible subjects must have PH documented as follows:

   1. Main Pulmonary Artery/Ascending Aorta (PA/A) diameter > 0.90 on clinically available CT scans within 12 months OR
   2. Main Pulmonary Artery diameter > 30.8mm on clinically available CT scans within 12 months OR
   3. outpatient echocardiography done within 6 months of enrollment demonstrating PA sys > 34 mmHg OR
   4. Mean Pulmonary Artery Pressure > 20 on Right Heart Catheterization done within 6 months of enrollment and when Veteran is clinically stable.
3. Eligible subjects must be dyspneic, as quantitated by a score of at least 20 on the baseline UCSD Shortness of Breath Questionnaire, assessed at the time of the baseline visit.
4. Treatment with at least one long-acting bronchodilator for at least 4 weeks, assessed at the time of the baseline visit by chart review and patient interview.
5. Age 35-89 Years
6. Women of childbearing potential must meet one of the following criteria for the previous three months AND must have a negative pregnancy test on the day of testing. If more than 36 hours since the participant's last pregnancy test, they will be tested again at the study visit.

   1. have been using a contraceptive measure (an intrauterine device (IUD), a contraceptive implant, oral contraceptives, barrier methods, or abstinence)
   2. have a male partner with a vasectomy
   3. have a tubal ligation procedure or a medical diagnosis (such as infertility) or therapies/procedures that precludes pregnancy (such as cancer treatments or endometrial ablation)
   4. are in a same-sex relationship
   5. have a male partner not capable of fathering children because of congenital anomalies, other surgery, or medical treatment
7. Women who are not considered to be of childbearing potential who have been surgically sterilized (for example: removal of ovaries or fallopian tubes, or hysterectomy) or are post-menopausal (no menstrual period for more than 6 months).

Exclusion Criteria:

1. Diagnosis of PH in the following subgroups of the updated WHO Clinical Classification:

   1. Group 1 (Idiopathic, heritable, drug- or toxin-induced, Pulmonary Arterial Hypertension associated with connective tissue disease, congenital heart disease)
   2. Group 2 (left atrial hypertension)
   3. Group 3 PH not attributable to COPD
   4. Group 4 (chronic thromboembolic PH) or other forms of PH not associated with primary lung disease.
2. Systemic hypotension in the ambulatory setting (at least 3 reproducible measurements of systolic BP <89 mmHg, recorded by a health care provider over 1 week).
3. Moderate or severe hepatic impairment (Child-Pugh B and C).
4. Severe renal insufficiency (GFR <30 ml/min/1.73 m2)
5. Echocardiography within 3 months showing greater than moderate aortic stenosis (aortic valve area <1.0 cm2), greater than moderate mitral regurgitation, or diastolic dysfunction (Any two of the following: Average E/e' >14, Septal e' velocity < 7 or lateral e' velocity <10, LA volume index > 34 ml/m2). LVEF < 50%. Any aortic or mitral valve replacement.
6. Any acute or chronic impairment (other than dyspnea) that limits ability to comply with the study requirements.
7. Current unstable angina, myocardial infarction or stroke within 6 months.
8. Requirement for nitrate therapy for any clinical indication.
9. Active prescription for a PDE-5 inhibitor or other pulmonary vasodilator other than oxygen as a PH treatment.
10. History of the following retinal disorders: retinitis pigmentosa, non-arteritic anterior ischemic optic neuropathy, or crowded optic disc noted on ophthalmology examinations recorded in CPRS.
11. Contraindications: PDE-5i allergy, penile anatomical deformations, sickle cell anemia, multiple myeloma, leukemia, bleeding disorders, active peptic ulcer disease, retinitis pigmentosa or other retinal disorders listed above. In accordance with 38 USC 7332, this information will be kept confidential and will not be disclosed in presentations, publications, or any other dissemination of the study results, or to anyone outside of the IRB-approved study team.
12. Use of any of the following: rifampin, systemic anti-fungal azole agents, protease inhibitors, phenobarbital, dilantin.
13. Pregnant, possibly pregnant by report, or if breastfeeding. If found to be pregnant at the study visit, the study visit will not be conducted.
14. Pulmonary veno-occlusive disease
15. Hypoxia (reproducible ambulatory SaO2 < 90% on supplemental oxygen at rest recorded by a health care provider over 1 week).
16. Diagnosis of Obstructive Sleep Apnea without a prescription for treatment.
17. Newly prescribed (less than 4 weeks duration) bronchodilator or diuretic therapy or new enrollment in pulmonary rehabilitation at the time of Baseline.
18. Students, VA employees, persons with impaired decision making, illiterate and non-English speakers, and terminally ill patients.
19. COPD or CHF exacerbation within the past 4 weeks.
20. On-going therapy with doxazosin.

Women of childbearing potential must have a documented negative pregnancy test and must be using adequate contraception during the study and for 9 months afterward. Monthly pregnancy tests will be done, and compliance with contraception use will be documented at the telephone and clinic visits. Should a female become pregnant at any time during the study, the study medication will be discontinued.

Doxazosin use will be defined as current active prescription and usage of Doxazosin or planned trial (pending prescription) of Doxazosin for treatment of benign prostatic hypertrophy, systemic hypertension, or other indication. A list of alpha-1 antagonists (ex. prazosin, doxazosin, tamulosin, terazosin, etc.) will be included in the patient study medication handout to prompt the patient to avoid any new usage of these drugs during the trial period. On-going therapy with doxazosin is an exclusion criterion due to greater risk of hypotension.

Ages: 35 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
severity of patient-reported dyspnea | 6 months
  Assessed by the University of California-San Diego Shortness of Breath Questionnaire (UCSD-SOBQ). Score range = 0-120 with higher scores indicating worse outcomes. Minimum score for inclusion in the study is 10.

SECONDARY OUTCOMES:
physical activity | 6 months
  assessed by objective average daily step count using actigraphy
clinically important deterioration | 6 months
  Defined as the presence or absence of at least one of the following: increase > 4U in the total health-related quality of life (St. George's Respiratory Questionnaire, SGRQ), decreased FEV1 of > 100mL, or moderate-severe acute exacerbation of COPD
functional exercise capacity | 6 months
  6 minute walk distance, defined as the distance walked in meters in 6 minutes

OTHER OUTCOMES:
Pulmonary artery to aorta diameter ratio | 6 months
  measured on low dose CT scan
Estimated PA systolic pressure in mm Hg | 6 months
  measured by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Sharon I Rounds, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (5):
- United States (5):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
1. Publications of results will be available to the public.
  2. The principal investigator will share de-identified datasets, statistics, and results collected from this proposal by depositing these data at the National Library of Medicine (NLM) PubMed Central website repository as this is a VA supported data repository. Additional documentation including metadata that will include information about the methodology and study procedures used to collect the data, details about code, definition of variables will also be included.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Above will be shared upon approval of the study.
Access Criteria: Individual participant data will be shared within one year of publication of results.